CLINICAL TRIAL: NCT03265457
Title: The Corneal Endothelial Cell Count in Eyes With Pseudoexfoliation Syndrome
Brief Title: The Endothelial Count in Pxf
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Asem, Principal investigator, Assiut University
Other Study IDs: PXF
Record Dates: First submitted 2017-08-26; First posted 2017-08-29 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Pseudoexfoliation Syndrome
MeSH Terms: conditions — Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient with pseudoexfoliation syndrome: The corneal Endothelial cell count will be measured by specular microscopy
  Interventions: Other: Specular microscopy
- Normal people at same age
  Interventions: Other: Specular microscopy

INTERVENTIONS:
Other: Specular microscopy — Comparison between corneal Endothelial count in patients with pseudoexfoliation syndrome and age matched group

SUMMARY:
Pseudoexfoliation Syndrome Is a common disorder in Egypt. IT is one of the common causes of coexisting cataract and glaucoma. It may be associated with a less than normal endothelial count.

DETAILED DESCRIPTION:
The corneal Endothelium is essential for the maintenance of normal corneal hydration, thickness, and transparency.

In patients with pseudoexfoliation syndrome , quantitative and qualitative morphological changes of the corneal endothelium have been demonstrated in specular and electron microscopic studies.

Specular microscopy is a non-invasive technique to access the structure and function of the corneal endothelium.

Our research question is to study Endothelial cell count in patients with pseudoexfoliation syndrome & compare it to age matched group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pseudoexfoliation syndrome

Exclusion Criteria:

* Patients with previous intra ocular surgeries.
* Patients with uveitis
* Patients with fuck's endothelial dystrophy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pseudoexfoliation syndrome
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between endothelial cell count in patients with Pseudoexfoliation syndrome and age matched controls. | One year
  The corneal Endothelial cell count in patients with pseudoexfoliation syndrome will be measured by the specular microscopy & compared with the normal endothelial count in people at the same group

REFERENCES:
- [Background] Miyake K, Matsuda M, Inaba M. Corneal endothelial changes in pseudoexfoliation syndrome. Am J Ophthalmol. 1989 Jul 15;108(1):49-52. doi: 10.1016/s0002-9394(14)73259-3. PMID 2750833